CLINICAL TRIAL: NCT02875730
Title: A Pilot Investigation Detecting Cryoablation Scar by 3D Late Gadolinium
Brief Title: A Pilot Investigation Detecting Cryoablation Scar by 3D Late Gadolinium Enhancement
Acronym: LAMDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aspire Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-044
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation; Cryoablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CMRI Pulse Sequence (Experimental): Patients will have late gadolinium cardiac magnetic resonance images of the individual pulmonary veins acquired with the standard and the cylindrical navigator preparatory pulse sequences for comparison.
  Interventions: Procedure: Pulse Sequence; Procedure: CMRI

INTERVENTIONS:
Procedure: Pulse Sequence — Cylindrical Navigator Preparatory Pulse Sequence
Procedure: CMRI — Cardiac Magnetic Resonance Imaging

SUMMARY:
This is a prospective trial investigating the effectiveness of a modified MRI preparatory pulse sequence to improve pulmonary vein isolation visualization.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women
* A diagnosis of symptomatic paroxysmal or recently persistent atrial fibrillation with a documented successful cardioversion within 4 months of the procedure
* Documented treatment failure or intolerance of at least 1 anti-arrhythmic medication used to control atrial fibrillation.

Exclusion Criteria:

* Contraindication to MRI, such as implanted incompatible metal prosthesis, or subject size exceeds bore or table limits
* Allergy to gadolinium-based contrast agent
* Previous atrial fibrillation ablation
* Renal dysfunction (estimated GFR <60 mL/min/1.73m2) within 6 months
* Unwilling to provide informed consent for this protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Blood Pool Corrected Signal Intensity | Through study completion, an average of 1 year
Imaging Failure Rate | Through study completion, an average of 1 year
Extent of Detected LGE Signal Correlate to the Respiratory Navigator Scheme | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's Health System, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No